CLINICAL TRIAL: NCT02576314
Title: Efficacy and Safety Study of Sofosbuvir Containing Regimens in Subjects With Chronic Hepatitis C Virus Genotype 3 Infection
Brief Title: Sofosbuvir Containing Regimens for the Treatment of Chronic HCV GT3 Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Humanity and Health Research Centre (Other)
Collaborators: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H&H_HCV G3 Study
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Chronic Hepatitis C Infection
MeSH Terms: interventions — Sofosbuvir; daclatasvir; ledipasvir, sofosbuvir drug combination; ledipasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sofosbuvir and Daclatasvir (Active Comparator): Participants will receive Sofosbuvir (SOF) 400 mg and Daclatasvir (DCV) 60 mg daily for 12 weeks.
  Interventions: Drug: sofosbuvir and daclatasvir
- Ledipasvir/sofosbuvir (Active Comparator): Participants will receive Ledipasvir/sofosbuvir (LDV/SOF) 90 mg/400 mg fixed dose combination (FDC) tablet daily for 12 weeks.
  Interventions: Drug: ledipasvir/sofosbuvir

INTERVENTIONS:
Drug: sofosbuvir and daclatasvir — Sofosbuvir (SOF) 400 mg tablet administered orally once daily. Daclatasvir (DCV) 60 mg tablet administered orally once daily.
  Other Names: Sovaldi®; PSI-7977; GS-7977; Daklinza®; BMS-790052
  Arms: Sofosbuvir and Daclatasvir
Drug: ledipasvir/sofosbuvir — Ledipasvir/sofosbuvir (LDV/SOF) 90 mg/400 mg fixed dose combination (FDC) tablet administered orally.
  once daily;
  Other Names: Harvoni®; GS-5885; GS-7977; PSI-7977
  Arms: Ledipasvir/sofosbuvir

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of Sofosbuvir containing regimens in treatment-naive or treatment-experienced patients with HCV genotype 3 infection.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years, with chronic genotype 3 HCV infection;
* Documented HCV treatment-naïve or treatment-experienced subjects who failed previous PEG+RBV regimen;
* HCV RNA > 10,000 IU/mL at Screening;
* Screening laboratory values within defined thresholds;
* Negative pregnancy test at baseline (females of childbearing potential only);
* Use of two effective contraception methods if female of childbearing potential or sexually active male.

Exclusion Criteria:

* Pregnant or nursing female;
* HIV infection or HBV infection (HBcAb and HBsAg positive);
* Hematologic or biochemical parameters at Screening outside the protocol-specified requirements;
* Active or recent history (≤ 1 year) of drug or alcohol abuse;
* Hepatocellular carcinoma or other malignancy (with exception of certain resolved skin cancers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-05; Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with sustained virologic response 12 weeks (SVR12) after discontinuation of therapy | Post treatment Week 12
  SVR12 is defined as HCV RNA < the lower limit of quantitation (LLOQ < 25 IU/mL) 12 weeks following the last dose of study medication
Incidence of adverse events leading to permanent discontinuation of study drug | Baseline up to Week 12

SECONDARY OUTCOMES:
Proportion of participants with unquantifiable HCV viral load at specified time points during and after treatment | Baseline up to Week 12
HCV RNA levels and change during and after treatment | Baseline up to Week 12
Treatment adherence | Baseline to Week 12
  To evaluate the proportion of patients adherent to therapy (both on-treatment adherence and treatment discontinuation)
Change in health related quality of life | Baseline to Week 24
  To evaluate the change in health-related quality of life during treatment

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, MD, Principal Investigator — Humanity and Health GI and Liver Centre
Locations (2):
- China (2):
  - Liver Fibrosis Diagnosis and Treatment Centre, 302 Hospital, Beijing, Beijing Municipality
  - Humanity and Health GI and Liver Centre, Hong Kong, Hong Kong